CLINICAL TRIAL: NCT05113043
Title: Research on Correlation Between Intestinal Microecology Imbalance and the Risk and Prognosis of Stroke in Young Adults
Brief Title: Correlation Between Intestinal Microecology Imbalance and Stroke in Young Adults
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, MD, PhD, Associate Clinical Professor, Shanghai 6th People's Hospital
Other Study IDs: 2021-KY-112 (K)
Record Dates: First submitted 2021-11-05; First posted 2021-11-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: ischemic stroke; hemorrhagic stroke; intestinal microecology; multi-omics analysis; prognosis
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faecal samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ischemic stroke: Young patients who suffered from acute ischemic stroke within 12 hours for the first time before entry into the study.
- Hemorrhagic stroke: Young patients who suffered from acute hemorrhagic stroke within 12 hours for the first time before entry into the study.
- Healthy Controls: Healthy young people

SUMMARY:
The relationship between the intestinal microecology and stroke has become a research hotspot in neurology field today. Maintaining the balance of the intestinal microbiota are expected to bring new breakthroughs for prevention and treatment of stroke. In recent years, stroke in young adults has an increasing incidence and a considerable socioeconomic impact because of high disability rate and health-care costs. So there is an urgent need to explore the role and mechanism of intestinal microecology imbalance in stroke, especially in the development and prognosis of stroke in young people. This study aims to use multi-omics technologies, including microbial diversity, metagenomics and metabonomics, to reveal the characteristics of intestinal flora in young stroke patients, identify biomarkers for predicting outcome after stroke and early detection of young people at high risk of stroke, and to further explore the role of gut-brain axis in the pathogenesis of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic or hemorrhagic stroke
* Admission within 12 hours
* Aged 18-45 years

Exclusion Criteria:

* History of neurological diseases, myocardial infarction, renal and hepatic abnormalities and metabolic diseases
* Combined with tumors, inflammatory bowel disease and other digestive system diseases
* Combined with serious life-threatening diseases or condition
* Any antibiotics, probiotics or prebiotic treatment within 3 months
* Deteriorate and die before collecting faecal samples

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young patients (18-45 years old) with ischemic or hemorrhagic stroke, who are admitted within 12 hours post-stroke are included. To avoid interfering factors, patients with existing prior neurological disease or known tumors, inflammatory bowel disease and other digestive system diseases, patients with serious life-threatening diseases or condition, patients under antibiotics, probiotics or prebiotic treatment within 3 months before stroke, and patients who deteriorate and die before collecting faecal samples are excluded. Clinical data are documented, including age, gender, types of stroke as evidenced by imaging examination and laboratory examination, etc.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale scores | 3 months
  0 = No symptoms; 1 = No significant disability. Able to carry out all usual activities, despite some symptoms; 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 = Moderate disability. Requires some help, but able to walk unassisted; 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 = Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Lixia Xue, M.D., Ph.D., Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, China